CLINICAL TRIAL: NCT05337254
Title: A Randomized, Open-Label, 5-Period Crossover Study to Evaluate the PK, Bioavailability, Safety, and Tolerability of Single Doses of STS101, DHE IM Injection and DHE Nasal Spray in Healthy Adult Subjects
Brief Title: A Study of the PK and Safety of Single Doses of STS101, DHE Injection and Nasal Spray in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Satsuma Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STS101-006
Record Dates: First submitted 2022-03-29; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Migraine; Migraine With Aura; Migraine Without Aura
Keywords: dihydroergotamine; dihydroergotamine mesylate; migraine
MeSH Terms: conditions — Migraine Disorders; Migraine with Aura; Migraine without Aura | interventions — Dihydroergotamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- STS101 5.2 mg (Experimental): STS101 (dihydroergotamine nasal powder), 5.2 mg
  Interventions: Drug: Dihydroergotamine
- STS101 7.0 mg (Experimental): STS101 (dihydroergotamine nasal powder), 7.0 mg
  Interventions: Drug: Dihydroergotamine
- STS101 8.6 mg (Experimental): STS101 (dihydroergotamine nasal powder), 8.6 mg
  Interventions: Drug: Dihydroergotamine
- DHE intramuscular injection (Active Comparator): Dihydroergotamine mesylate
  Interventions: Drug: Dihydroergotamine
- DHE nasal spray (Active Comparator): Dihydroergotamine mesylate
  Interventions: Drug: Dihydroergotamine

INTERVENTIONS:
Drug: Dihydroergotamine — Dihydroergotamine intranasal powder
  Other Names: Dihydroergotamine Mesylate
  Arms: STS101 5.2 mg; STS101 7.0 mg; STS101 8.6 mg
Drug: Dihydroergotamine — Dihydroergotamine intramuscular injection
  Other Names: Dihydroergotamine Mesylate
  Arms: DHE intramuscular injection
Drug: Dihydroergotamine — Dihydroergotamine intranasal spray
  Other Names: Dihydroergotamine Mesylate
  Arms: DHE nasal spray

SUMMARY:
Single-center, single-dose, open-label, 5-period crossover (in each part), pharmacokinetic and safety study.

DETAILED DESCRIPTION:
36 subjects received a single dose of STS101, 1.0 mg DHE mesylate IM injection, and 2 mg DHE mesylate nasal spray in a randomized, 5-period crossover manner.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 50 years of age at the time of enrollment.
* Signed the informed consent document.
* Subject judged to be healthy by a qualified physician

Exclusion Criteria:

* Abnormal physical findings of clinical significance at the screening examination
* Significant abnormal laboratory values at the Screening Visit.
* Clinically significant symptoms or conditions that may have placed the subject at an unacceptable risk as a participant in the trial, or that may have interfered with the absorption, distribution, metabolism or excretion of the IMP.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-06-04 (Actual); Study Completion 2021-06-04 (Actual)

PRIMARY OUTCOMES:
DHE Relative Bioavailability | Pre-dose through 48 hours Post-Dose
  The relative bioavailability of STS101 5.2, 7.0, and 8.6 mg (test treatments) to 1.0 mg DHE mesylate IM injection (reference treatment) and to 2.0 mg DHE mesylate IN spray (reference treatment) was assessed on the basis of dose-corrected Cmax.
DHE Comparative Bioavailability | Pre-dose through 48 hours Post-Dose
  The comparative bioavailability STS101 5.2, 7.0, and 8.6 mg (test treatments) to 1.0 mg DHE mesylate IM injection (reference treatment) and to 2.0 mg DHE mesylate IN spray (reference treatment) was assessed on the basis of Cmax .

SECONDARY OUTCOMES:
Serious Adverse Events | Pre-dose through 48 hours Post-Dose
  To assess the safety profile through examination of serious adverse events of single doses of STS101; 1 mg DHE administered by intramuscular injection, and 2 mg DHE administered as nasal spray
Treatment-Related Adverse Events | Pre-dose through 48 hours Post-Dose
  To assess the safety profile through examination of treatment-related adverse events of single doses of STS101; 1 mg DHE administered by intramuscular injection, and 2 mg DHE administered as nasal spray

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Levy, MD, Principal Investigator — Quotient Sciences Miami Inc
Locations (1):
- Quotient Sciences Miami Inc., Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lipton RB, Albrecht D, Bermudez M, Hu J, Hussey E, Levy J. A randomized, open-label, 5-period crossover study evaluating the pharmacokinetics and safety of a single dose of intranasal dihydroergotamine (DHE) powder (STS101), intramuscular DHE mesylate, and liquid nasal spray DHE in healthy adults. Headache. 2024 Mar;64(3):266-275. doi: 10.1111/head.14685. Epub 2024 Feb 27. PMID 38413540